CLINICAL TRIAL: NCT00064428
Title: An International Randomized Study Evaluating the Efficacy and Safety of Fondaparinux Versus Control Therapy in a Broad Range of Patients With ST Segment Elevation Acute Myocardial Infarction.
Brief Title: OASIS-6 : The Safety and Efficacy of Fondaparinux Versus Control Therapy in Patients With ST Segment Elevation Acute Myocardial Infarction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 103413; NCT01352156 (obsolete NCT alias)
Record Dates: First submitted 2003-07-08; First posted 2003-10-17 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Thromboembolism
Keywords: ST-segment elevation myocardial infarction; fondaparinux; Acute Myocardial Infarction; acute coronary syndrome
MeSH Terms: conditions — Thromboembolism; ST Elevation Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fondaparinux - UFH not indicated (Experimental): Subjects with no indication for UFH therapy: 2.5mg od, sc, (1st dose IV) x 8 days or discharge
  Interventions: Drug: fondaparinux - UFH not indicated
- Control - UFH not indicated (Placebo Comparator): Subjects with no indication for UFH therapy: Fondaparinux-placebo od, sc (1st dose IV) x 8 days or discharge
  Interventions: Other: Control - UFH not indicated
- Fondaparinux - UFH indicated (Experimental): Subjects indicated for UFH: 2.5mg od, sc (1st dose IV) x 8 days or discharge + UFH-placebo IV bolus + 24-48 hr infusion
  Interventions: Drug: Fondaparinux - UFH indicated
- Control - unfractionated heparin (Active Comparator): Subjects indicated for UFH: UFH IV bolus +12 IU/kg/hr infusion x 24-48 hr + fondaparinux-placebo od, sc (1st dose IV) x 8 days or discharge
  Interventions: Drug: Control - UFH

INTERVENTIONS:
Drug: fondaparinux - UFH not indicated — 2.5mg od, sc (1st dose IV) x 8 days or discharge
  Arms: Fondaparinux - UFH not indicated
Other: Control - UFH not indicated — Fondaparinux-placebo od, sc (1st dose IV) x 8 days or discharge
  Arms: Control - UFH not indicated
Drug: Fondaparinux - UFH indicated — 2.5mg od, sc (1st dose IV) x 8 days or discharge + UFH-placebo IV bolus x 24-48 hr infusion
  Arms: Fondaparinux - UFH indicated
Drug: Control - UFH — UFH IV bolus +12 IU/kg/hr infusion x 24-48 hr + fondaparinux-placebo od, sc (1st dose IV) x 8 days or discharge
  Arms: Control - unfractionated heparin

SUMMARY:
This is a randomized, double blindcontrolled, parallel group, multi-center, multinational study of fondaparinux vs. control in patients with STEMI (ST segment myocardial infarction) randomized within 24 hours of the onset of symptoms.

DETAILED DESCRIPTION:
This is a randomized, double blind, controlled, parallel group, multi-center, multinational study of fondaparinux vs. control in patients with STEMI randomized within 24 hours of the onset of symptoms. Patients with confirmed STEMI were assigned into one of the following strata, based on local preference:

Stratum 1: No indication for UFH; it is generally accepted that patients receiving streptokinase or those not receiving a thrombolytic agent were assigned to this stratum.

Stratum 2: Indication for UFH; it is generally accepted that patients receiving a fibrin-specific agent (such as alteplase, reteplase or tenecteplase) or those undergoing primary PCI were assigned to this stratum.

Patients who were ineligible for fibrinolysis (e.g. because of late presentation or absolute contra-indication for reperfusion therapy) may fall into either stratum 1 or stratum 2 at investigator's discretion. Following allocation to one of the strata, patients were randomized to fondaparinux or control treatment. Control treatment was dependent on whether the patient was assigned to stratum 1 or stratum 2:

Stratum 1: fondaparinux sc* versus fondaparinux-placebo sc for 8 days or until hospital discharge, whichever was earlier.

Stratum 2: fondaparinux sc* for 8 days or until hospital discharge, whichever was earlier and UFH-placebo for 24 to 48 hrs (or single bolus injection immediately prior to procedure in case of primary PCI) versus UFH for 24 to 48 hrs (or single bolus injection immediately prior to procedure in case of primary PCI) and fondaparinux-placebo for 8 days or until hospital discharge, whichever was earlier.

(*First dose intravenous bolus) Patients were followed up for 6 months

ELIGIBILITY:
Inclusion Criteria:

* Subjects who presented or were admitted to hospital with:

  1. Signs and symptoms of AMI
  2. Were able to randomize within 12 hours of symptom onset; and-
  3. Had definite ECG changes indicating STEMI: persistent ST-elevation (≥0.2mV in two contiguous precordial leads, or ≥0.1mV in at least two limb leads), or new left bundle branch block, or ECG changes indicating true posterior MI.
* Written informed consent
* Able to be randomized within 24 hours of symptom onset

Exclusion Criteria:

* Age <21 years.
* Was currently receiving an oral anticoagulant agent with an INR >1.8.
* Had any contraindication to anticoagulation therapy such as high risk of bleeding or active bleeding.
* Had hemorrhagic stroke within the last 12 months.
* Had an indication for anticoagulation other than ACS.
* Pregnant women or women of child-bearing potential who were not using an effective method of contraception.
* Had a co-morbid condition with a life-expectancy <6 months.
* Previous enrollment in one of the fondaparinux ACS trials.
* Participation in another pharmacotherapeutic study within the prior 30 days or was currently receiving an experimental pharmacological agent.
* Had a known allergy to heparin or fondaparinux.
* Had severe renal insufficiency (i.e. serum creatinine ≥3mg/dL or ≥265μmol/L).
* Had >5000IU UFH administered prior to randomization.
* Had LMWH administered prior to randomization.
* Subject had pre-randomization revascularization (PCI) for the index event.
* Subject had pre-randomization rescue PCI.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12092 (Actual)
Dates: Start 2003-08; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Death or recurrent myocardial infarction | up to day 30
  the first occurrence of any component of death (all-cause mortality) or recurrent myocardial infarction
Severe hemorrhage | up to Day 9
  Severe hemorrhage (modified TIMI criteria)

SECONDARY OUTCOMES:
Death or recurrent myocardial infarction | up to Day 9, 90 and 180
  The first occurrence of any component of the composite of death (all-cause mortality) or recurrent myocardial infarction
Death, recurrent myocardial infarction or refractory ischemia | up to Day 9, 30, 90 and 180
  The first occurrence of any component of the composite of death (all-cause mortality), recurrent myocardial infarction or refractory ischemia

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Yusuf S, Mehta SR, Chrolavicius S, Afzal R, Pogue J, Granger CB, Budaj A, Peters RJ, Bassand JP, Wallentin L, Joyner C, Fox KA; OASIS-6 Trial Group. Effects of fondaparinux on mortality and reinfarction in patients with acute ST-segment elevation myocardial infarction: the OASIS-6 randomized trial. JAMA. 2006 Apr 5;295(13):1519-30. doi: 10.1001/jama.295.13.joc60038. Epub 2006 Mar 14. PMID 16537725
- [Derived] Diaz R, Goyal A, Mehta SR, Afzal R, Xavier D, Pais P, Chrolavicius S, Zhu J, Kazmi K, Liu L, Budaj A, Zubaid M, Avezum A, Ruda M, Yusuf S. Glucose-insulin-potassium therapy in patients with ST-segment elevation myocardial infarction. JAMA. 2007 Nov 28;298(20):2399-405. doi: 10.1001/jama.298.20.2399. PMID 18042917
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 103413 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 103413 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 103413 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 103413 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 103413 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 103413 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 103413 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register